CLINICAL TRIAL: NCT06705335
Title: Convertases and Pancreatic Cancer. New Therapeutic and Prognostic Approach: Cohort of Patients Treated for Pancreatic Adenocarcinoma (CONVERCAP)
Brief Title: Convertases and Pancreatic Cancer: Cohort of Patients Treated for Pancreatic Adenocarcinoma
Acronym: CONVERCAP
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB 2024-01; 2024-A01797-40 (Other: ID-CRB)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Pancreas Cancer
Keywords: Convertases
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pancreas or metastases tumor sample Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CONVERCAP patients: The tumour sample (primary tumour or metastasis) will be taken either during a standard biopsy or during pancreatic or metastasis standard surgery.
  Biopsy sampling of metastases is only authorised if the primary histological diagnosis of pancreatic adenocarcinoma has already been proven. If the patient has undergone a biopsy for diagnostic purposes, he/she cannot be included in the study.
  The blood sample will be taken on the same day as the tumour sample.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — On the same day as the tumour sample is taken (biopsy or surgery), a blood sample of approximately 15 to 20 mL is taken in EDTA-free tubes.

SUMMARY:
This is a prospective, single-centre, observational study. The analysis of samples of pancreatic tumours and/or metastases taken during biopsy or surgery will lead to the determination of the level of expression of convertases in patients with pancreatic cancer and could be used as an additional prognostic means reinforcing those currently used.

DETAILED DESCRIPTION:
After checking the inclusion criteria and signing the consent form, patients will be pre-selected for the study.

A tumour sample (primary tumour or metastasis) will be taken either during a biopsy or during pancreatic or metastasis surgery.

A blood sample will be taken on the same day as the tumour sample. The inclusion visit will be carried out by the investigating physician and will correspond to the visit when the results of the biopsy or surgery are reported.

Inclusion of the patient will be possible if the tumour sample has been taken, is available, contributory and malignant (diagnosis or confirmation of pancreatic adenocarcinoma) and if the blood sample has been taken and is available.

The patient will be considered to have failed pre-selection if

* the tumour sample has not been taken or is not available, or
* the tumour sample/histological result is non-contributory, or
* the histological result is benign, or
* the blood sample was not taken or is not available, or
* the patient refuses to continue the study, or
* the patient has withdrawn consent, or
* any other reason preventing inclusion of the patient. Included patients will be treated and followed as usual, with standard radiological follow-up.

For two years after inclusion, the tumour status (first progression) and vital status of the patient (alive, dead or lost to follow-up at the date of the visit) will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Pancreatic adenocarcinoma (suspected on radiological assessment or histologically proven):

   1. Indication for biopsy of metastasis(es) performed as part of standard care for patients who already have a histologically confirmed diagnosis of pancreatic cancer.
   2. Indication for pancreatic surgery or metastasis(es) carried out as part of standard care for patients with a suspicion of pancreatic cancer on radiological assessment or who already have a confirmed histological diagnosis of pancreatic cancer.
3. Whatever the stage of the disease.
4. Whatever the type of treatment proposed (systemic, surgery, radiotherapy, etc.).
5. Patient who has never received systemic treatment or advanced radiotherapy.
6. WHO 0-1-2.
7. Life expectancy > 3 months.
8. Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).
9. Patient affiliated to a social security scheme in compliance with Article 1121-11 of the French Public Health Code.

Exclusion Criteria:

1. Indication for biopsy for primary diagnosis of pancreatic cancer
2. No indication for treatment of pancreatic cancer.
3. Adjuvant/neoadjuvant chemotherapy completed less than 6 months ago in the case of patients with recurrent disease.
4. Patient already included in the study.
5. Geographical, social or psychological factors rendering the patient unable to undergo study monitoring and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pancreatic adenocarcinoma (suspected on radiological assessment or histologically proven), whatever the stage of the disease ot the type of treatment proposed (systemic, surgery, radiotherapy, etc.), undergoing a biopsy or a surgery to collect tumor and blood samples.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficients between level of expression of various convertases on the tumor and immune infiltrate | Inclusion, Day 1
  The level of expression of convertase proteins and their substrates (VEGF-C, IGF-1) will be determined on tumor samples at inclusion (healthy tissues, primary cancers and metastases), using qRT-PCR, western blot, ELISA, FACs and/or immunofluorescence as methodology and will be correlated with the following immune parameters, determined by immunofluorescence (including but not limited to): CD8, CD4, NK,Tregs, Macrophages
  The analysis will assess the correlation between the expression of various convertases on the tumor and immune parameters using Pearson's correlation coefficient for normally distributed variables, or Spearman's correlation coefficient for non-normally distributed variables. The correlation coefficient ranges from -1 to 1: a value closer to 1 indicates a strong positive association, a value closer to -1 indicates a strong negative association, and a value closer to 0 indicates no association.

SECONDARY OUTCOMES:
Correlation coefficients between level of expression of various convertases determined at plasma level and immune infiltrate | Inclusion, Day 1
  The level of expression of convertase proteins will be determined at plasma level at inclusion, using qRT-PCR, western blot, ELISA, FACs and/or immunofluorescence as methodology and will be correlated with the following immune parameters, determined by immunofluorescence (including but not limited to): CD8, CD4, NK,Tregs, Macrophages.
  The analysis will assess the correlation between the expression of various convertases on plasma and immune parameters using Pearson's correlation coefficient for normally distributed variables, or Spearman's correlation coefficient for non-normally distributed variables. The correlation coefficient ranges from -1 to 1: a value closer to 1 indicates a strong positive association, a value closer to -1 indicates a strong negative association, and a value closer to 0 indicates no association.

CONTACTS AND LOCATIONS:
Overall Officials: Simon PERNOT, Dr, Principal Investigator — Institut Bergonié